CLINICAL TRIAL: NCT06310616
Title: A Phase 1, Single-center, Open-label Study to Evaluate the Pharmacokinetics of Oral Contraceptive Containing Norethindrone and Ethinyl Estradiol (Loestrin) When Co-administered With VH4524184 in Healthy Adult Female Participants
Brief Title: A Study to Investigate the Potential Drug-Drug Interaction Between VH4524184 and Oral Contraceptive (Loestrin) in Healthy Adult Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 219888
Record Dates: First submitted 2024-03-01; First posted 2024-03-15 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections
Keywords: HIV; Oral contraceptive; Pharmacokinetic; Ethinyl estradiol; Norethindrone acetate; Potential drug-drug interaction; Healthy adult female participants
MeSH Terms: conditions — HIV Infections | interventions — norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Loestrin + VH4524184 (Experimental): Eligible participants entering a run-in period of 21 days (Days -28 through -8) will receive Loestrin (EE and NEA) to stabilize on the combined OCs containing EE and NEA to synchronize the menstrual cycles of multiple participants. Participants completing the run-in period will enter Treatment Period 1 and will be administered Loestrin once daily from Days 1 to 10. On Day 11, participants will enter Treatment Period 2 and will be administered Loestrin + VH4524184 once daily from Days 11 to 20.
  Interventions: Drug: VH4524184; Drug: Loestrin

INTERVENTIONS:
Drug: VH4524184 — VH4524184 will be administered.
Drug: Loestrin — Loestrin will be administered.

SUMMARY:
This study aims to assess any impact of VH4524184 on the pharmacokinetic (PK) profile of an ethinyl estradiol (EE) and norethindrone acetate (NEA) containing oral contraceptive (OC) administered to healthy adult female participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants 18 to 45 years of age
* POCBP with intact ovarian function by medical history and history of regular menstrual cycles for the past 12
* Body weight greater than or equal to (≥) 45 kilograms (kg) and Body mass index (BMI) within the range of 18.5 to 32.0 kg/m2
* Female participants of childbearing potential must use approved highly effective non-hormonal forms of birth control.
* Capable of giving signed informed consent.

Exclusion Criteria:

* History or presence of clinical condition or disorder that could be capable of significantly altering the absorption, metabolism, or elimination of drugs.
* Lymphoma, leukemia, or any malignancy within the past 5 years with some exceptions
* Breast cancer or in remission within the past 10 years.
* Current or chronic history of liver disease or known hepatic or biliary abnormalities with some exceptions.
* Any personal and/or family history of thrombophilia or blood clots
* Medical history of cardiac arrhythmias or cardiac disease or a family and personal history of long QT syndrome.
* History of seizure(s).
* Any known or suspected pre-existing psychiatric condition, including depression, anxiety, and/or insomnia/sleep disturbances.
* Subjects with history of drug hypersensitivity, delayed-type hypersensitivity, or severe hypersensitivity reactions, as well as history of sensitivity to the study interventions will be excluded.
* Participant is mentally or legally incapacitated.

Prior/Concomitant Therapy

• Any warnings and contraindications that apply based on Loestrin prescribing information.

Prior/Concurrent Clinical Study Experience

* Exposure to more than 4 new investigational products (including long-acting investigational products) within 12 months prior to the first dosing day.
* Current enrollment or past participation in another investigational study in which an investigational intervention was administered within the last 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer) before signing of consent (or screening) any other clinical study.
* Participant has donated or lost blood (>500 millilitres (mL)) or blood products within 2 months (56-day period) prior to Day -1 admission or has donated plasma within 30 days prior to first OC administration.
* Current enrollment or past participation in this clinical study. Unwillingness or inability to follow the procedures outlined in the protocol.
* Positive Human immunodeficiency virus 1 (HIV-1) antibody test.
* Pregnant at screening) or lactating.
* POCBP who are unwilling or unable to use an appropriate non-hormonal method of highly effective contraception from at least Day 1 of Treatment Period 1 until 14 days after the last dose of VH4524184.
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >7 units for females. One unit is equivalent to 8 grams (g) of alcohol: a half-pint (~240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits.
* Regular use of known drugs of abuse.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female participants of childbearing potential (POCBP)
Enrollment: 26 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC) from time zero (pre-dose) to the end of the dosing interval at steady state (AUC0-Tau, ss) of EE and NEA without coadministration with VH4524184 | On Day 10
  Blood samples will be collected at indicated timepoint for plasma EE and NEA PK analysis.
AUC0-Tau, ss of EE and NEA with coadministration with VH4524184 | On Day 20
  Blood samples will be collected at indicated timepoint for plasma EE and NEA PK analysis.
Maximum plasma concentration (Cmax) for EE and NEA without coadministration with VH4524184 | On Day 10
  Blood samples will be collected at indicated timepoint for plasma EE and NEA PK analysis.
Cmax for EE and NEA with coadministration with VH4524184 | On Day 20
  Blood samples will be collected at indicated timepoint for plasma EE and NEA PK analysis.

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) and severity of AEs | From Day -28 (Run-In-Period) up to approximately 2 months (Day 28 +/- 3 days)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Number of participants with AEs leading to discontinuation of study intervention | Throughout the study treatment period (from Day -28 up to Day 20)
Change from baseline of liver panel laboratory parameters: Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (ASP) (International units per liter) | Baseline (Day -28) up to Day 21
Change from baseline of liver panel laboratory parameters: Total bilirubin, Direct bilirubin (Micromoles per liter [umol/L]) | Baseline (Day -28) up to Day 21
Change from baseline of liver panel laboratory parameters: International normalized ratio (INR) (Ratio) | Baseline (Day -28) up to Day 21
Number of participants with maximum toxicity grade increase from baseline of liver panel laboratory parameters: ALT, AST, alkaline phosphatase, total bilirubin, Direct bilirubin, and INR | Baseline (Day -28) up to Day 21
Maximum plasma concentration at steady state (Cmax,ss) for VH4524184 | On Day 20
  Blood samples will be collected at indicated timepoint for plasma VH4524184 PK analysis.
Time to maximum concentration at steady state (Tmax, ss) during dosing interval for VH4524184 | On Day 20
  Blood samples will be collected at indicated timepoint for plasma VH4524184 PK analysis.
Area under the concentration-time curve from time zero(pre-dose) to the end of the dosing interval at steady state (AUC0-Tau, ss) for VH4524184 | On Day 20
  Blood samples will be collected at indicated timepoint for plasma VH4524184 PK analysis.
Trough concentration prior to the next dose (Ctrough) for VH4524184 | On Day 12, Day 16, and Day 20
  Blood samples will be collected at indicated timepoints for plasma VH4524184 PK analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/